CLINICAL TRIAL: NCT01792089
Title: Measure of Intestinal Lipogenesis in Healthy Volunteers and Obese Subjects Before and After Gastroplasty: Modulation by Glucose and Fructose
Brief Title: Fructose-induced Intestinal de Novo Lipogenesis
Acronym: FIDNL
Status: Completed | Type: Observational
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, Professor, University of Lausanne
Other Study IDs: 193/11
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Obesity
Keywords: de novo lipogenesis; fructose; roux-en-Y gastric bypass; post-prandial triglycerides
MeSH Terms: conditions — Obesity | interventions — CD36 Antigens; Proteins; Whey Proteins

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- non-obese healthy subjects: subjects with BMI<25 and no known disease
  Interventions: Other: fat+protein meal; Other: Fat + protein + 13C fructose meal; Other: Fat+protein+13C fructose+glucose meal; Other: 13C Fat + whey protein; Other: 13C Fat + whey protein + glucose+ glucose meal
- post-gastric bypass: post-obese subjects 12-48 months after Roux-en-Y gastric bypass
  Interventions: Other: fat+protein meal; Other: Fat + protein + 13C fructose meal; Other: 13C Fat + whey protein + glucose+ glucose meal
- matched control subjects: Nonobese, healthy subjects of similar age, weight, and gender ratio, than post-bypass subjects
  Interventions: Other: fat+protein meal; Other: Fat + protein + 13C fructose meal; Other: 13C Fat + whey protein + glucose+ glucose meal

INTERVENTIONS:
Other: fat+protein meal — cream+ whey protein
Other: Fat + protein + 13C fructose meal — cream+ whey protein +13C fructose
Other: Fat+protein+13C fructose+glucose meal — Cream + whey protein + glucose:13C fructose mixture
  Groups: non-obese healthy subjects
Other: 13C Fat + whey protein — cream labelled with 13C palmitate + whey protein
  Groups: non-obese healthy subjects
Other: 13C Fat + whey protein + glucose+ glucose meal — cream labelled with 13C palmitate + whey protein + glucose:fructose mixture

SUMMARY:
8 healthy volunteers, 8 pre-bypass obese subjects, 8 subjects between 12-18 months post-bypass, and 8 subjects matched to the post-bypass patients will be studied in two sub-studies Sub-study 1) after ingestion of two or three different of the following test-meals: A)cream and whey protein B)cream, whey protein and fructose + 13C6 fructose C)test meal with cream, whey protein, fructose and glucose + 13C6 fructose Their intestinal de novo lipogenesis will be estimated by measuring 13C-palmitate on triglyceride-rich lipoprotein particles associated with apoB48 in blood Sub-study 2) after ingestion of two or three different of the following test-meals: A)cream labelled with 13C6 palmitic acid and whey protein B))cream labelled with 13C6 palmitic acid, whey protein, fructose and glucose

Their intestinal de novo lipogenesis will be estimated by measuring 13C-palmitate on triglyceride-rich lipoprotein particles associated with apoB48 in blood in sub-study 1

Their exogenous lipid absorption kinetics will be assessed by measuring 13C palmitate on triglyceride-rich lipoprotein particles associated with apoB48 in sub-study 2

ELIGIBILITY:
Inclusion Criteria:

* age 18-50 years
* sex male or female
* less than 2 kg body weight change over the past 3 months subjects

Exclusion Criteria:

* antidiabetic and hypolipemic drugs
* alcohol consumption >20g/day
* severe eating disorders
* severe psychological problems
* vegetarian diet or other specific diet
* consumption of illicit substances
* pregnancy
* weight gain or weight loss > 1 kg in the last 3 months

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 8 non-obese healthy male and female subjects with BMI <25 8 obese male and female subjects with BMI> 35 8 post-gastric bypass male and female subjects 8 healthy subjects matched to post-gastric bypass subjects for age, gender and weight
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Intestinal de novo lipogenesis (sub-study 1) | 0-8-hour post-prandial
  Measurement of total TG and 13C palmitate in chylomicrons: The sf >20 fraction of post-prandial blood samples will be prepared, and non-chylomicrons, apoB100-containing lipoprotein will be removes by immuno-affinity chromatography using a specific anti-apoB100 antibody
Postprandial exogenous, labelled palmitate concentration (sub-study 2) | 0-8-hour post-prandial
  Measurement of total TG and 13C palmitate in chylomicrons of sf >20 fraction of post-prandial blood samples will be prepared,

SECONDARY OUTCOMES:
post-prandial triglyceride profile (sub-studies 1 and 2 | 0-8 hour post-prandial
  Triglyceride will be measured in the chylomicron, VLDL, LDL and HDL fractions of post-prandial blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Theytaz F, de Giorgi S, Hodson L, Stefanoni N, Rey V, Schneiter P, Giusti V, Tappy L. Metabolic fate of fructose ingested with and without glucose in a mixed meal. Nutrients. 2014 Jul 15;6(7):2632-49. doi: 10.3390/nu6072632. PMID 25029210